CLINICAL TRIAL: NCT05962164
Title: The Acute and Chronic Benefits of Passive Heat Therapy for People With COPD
Brief Title: Passive Heat Therapy for People With COPD
Acronym: COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Lung Association (Industry)
Responsible Party: Principal Investigator, Neil Eves, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H21-01868
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: COPD; Cardiovascular Diseases
Keywords: Passive Heat Therapy; Pulmonary Rehabilitation; Cardiovascular Health
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Parallel 2-Arm Randomized Control Trial
Who Masked: Outcomes Assessor
Masking Description: Blinding of the participant to the condition (heat therapy or sham) is not possible. Data that needs to be analyzed (i.e. ultrasound videos for blood flow and FMD) will be coded by a team member that is not involved in data collection or analysis. The outcomes assessor will be blind to the participant, condition and time point of the file. Breaking of the code will only occur when all data analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive Heat Therapy (Experimental): Patients with COPD assigned to passive heat therapy will have their lower legs immersed in a circulating hot water (~42°C) footbath for 45 min per session.
  Interventions: Behavioral: Passive Heat Therapy
- Sham Immersion (Sham Comparator): Patients with COPD assigned to the sham condition will have their lower legs immersed in a circulating thermoneutral (~36°C) footbath for 45 min per session.
  Interventions: Behavioral: Sham Immersion

INTERVENTIONS:
Behavioral: Passive Heat Therapy — The intervention will consist of 6 weeks of repeated (3x/week) 45-min lower-leg immersions.
  Other Names: Lower-leg Hot Water Immersion; Footbath
  Arms: Passive Heat Therapy
Behavioral: Sham Immersion — The sham intervention will consist of 6 weeks of repeated (3x/week) 45-min lower-leg immersions.
  Arms: Sham Immersion

SUMMARY:
People with Chronic Obstructive Pulmonary Disease (COPD) often develop high blood pressure and heart disease due to their sedentary lifestyle and difficulty exercising. The investigators will test if heating can mimic the health benefits of exercise by monitoring the increase in leg blood-flow using ultrasound during a 45-minute hot-water footbath. The patients will then undergo 6-weeks of hot-water footbaths to examine whether the changes to blood-flow lead to improvements in blood pressure and other indicators of heart disease risk.

DETAILED DESCRIPTION:
People with COPD are at higher risk of developing cardiovascular disease (CVD). While exercise training is a potent therapy for CVD, people with COPD have a low tolerance for exercise due to dyspnea and premature muscle fatigue. Thus, there is a need to develop more effective strategies to improve CVD risk in people with COPD. A novel way to reduce blood pressure and enhance arterial health is with passive heat therapy (PHT). An acute 45-min bout of lower limb hot-water immersion has been shown to increase leg blood flow and reduce blood pressure in healthy older adults, suggesting that PHT could have similar hypotensive and anti-atherosclerotic effects as exercise. Augmenting leg blood flow with PHT may also have functional benefits by reducing peripheral muscle fatigue and improving exercise tolerance. No study to date has looked at the acute and chronic hemodynamic and vascular responses to PHT in people with COPD, nor whether it can acutely or chronically improve exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking individuals
* >40 years of age
* Stable (exacerbation free for >6 weeks), moderate-to-severe COPD (post bronchodilator FEV1/FVC <lower limit of normal and FEV1 z-score <2.51)

Exclusion Criteria:

* Performing structured exercise training (i.e. pulmonary rehabilitation)
* Have advanced cardiac or cerebrovascular disease (i.e. a history of heart failure, previous stroke or myocardial infarction)
* Have uncontrolled hypertension (>160/95 mmHg at rest)
* Have hypotension (<110/60 mmHg)
* Are taking Beta Blockers
* Regularly (>1/week) have hot baths (>30 min) or use a hot tub or sauna.

Exclusion Criteria for exercise outcomes:

* Have resting blood pressure > 150/95 mmHg
* On supplemental oxygen for hypoxemia.
* Musculoskeletal pain that limits their ability to perform stationary cycling.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean 24-hour ambulatory blood pressure following chronic passive heat therapy | 6 weeks
  The change in 24-hour ambulatory systolic, diastolic and mean arterial blood pressure from baseline to post intervention.

SECONDARY OUTCOMES:
Flow mediated dilation of the superficial femoral artery following chronic passive heat therapy. | 6 weeks
  The change in the percent dilation of the superficial femoral artery (measured using ultrasound) in response to reactive hyperemia (from a 5-min supra-systolic occlusion) from baseline to post intervention.
Arterial stiffness following chronic passive heat therapy | 6 weeks
  The change in pulse wave velocity (m/s) measured by applanation tonometry from baseline to post intervention.
Exercise tolerance following chronic passive heat therapy | 6 weeks
  The change in constant load exercise time (seconds) at 75% of peak power from baseline to post intervention.
The acute changes in leg blood flow from a single bout of passive heat therapy | During procedure: 60-minutes
  Superficial femoral artery blood flow (mL/min) will be measured by duplex ultrasound. Measurements will be taken every 15-min throughout immersion until 15-min following the first session of passive heat therapy or Sham treatment.
The acute changes in superficial femoral artery shear stress from a single bout of passive heat therapy | During procedure: 60-minutes
  Superficial femoral artery shear stress (1/s) patterns will be measured by duplex ultrasound. Measurements will be taken every 15-min throughout immersion until 15-min following the first session of passive heat therapy or Sham treatment.

OTHER OUTCOMES:
The acute change in exercise tolerance following a single bout of PHT vs. the change with sham treatment | ~48 hours
  Constant load exercise time to exhaustion (seconds) at 75% of Peak Power will be completed at baseline and 15-min after PHT or Sham Immersion. The change in post-PHT time to exhaustion from the baseline exercise trial will be compared with the change in post-sham time to exhaustion from the baseline exercise trial.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Eves, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No